CLINICAL TRIAL: NCT05571280
Title: Maternal and Child Interventions Against Chronic Malnutrition in Angola. A Cluster-randomized Cost-effectiveness Community-based Study.
Brief Title: Community-based, Controlled, Open-label, Cluster-randomized Trial for the Reduction of Chronic Malnutrition in Children Under Two Years of Age, With Three Intervention Arms Grouped by Clusters, in Two Provinces in Southern Angola, Huíla and Cunene.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Carlos III Health Institute (Other Government); Action Contre la Faim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MuCCUA
Record Dates: First submitted 2022-09-16; First posted 2022-10-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Intervention (Experimental): The Standard package includes a series of actions carried out by the Community and Health Development Agents (ADECOS), who improves access to primary health care practices and promotes well-being behaviors at community levels. ADECOS has the potential to facilitate improvements in the health state and quality of life in rural communities. Activities performed by ADECOS can be grouped into two blocks:
  * Health awareness-raising, and promotion activities at the community level (against malnutrition and promoting adequate nutrition).
  * Preventive community activities involving the promotion of treatment against malnutrition at the community level and direct referral to local health facilities when necessary.
  Interventions: Behavioral: Standard intervention
- Standard Intervention plus nutritional supplementation (Standard+NUT Arm) (Active Comparator): In addition to the services performed by the ADECOS, it is included a supply of complementary food rations (individual + family) at the relative level, being:
  * One individual portion composed by nutritional lipid supplements in small quantities (SQ-LNS)
  * One complementary family portion composed by local foods.
  Interventions: Dietary Supplement: Nutritional Supplementation
- Standard Intervention plus money transfers (Standard+TM Arm) (Experimental): In addition to the services performed by the ADECOS, it will be delivered a total of 14,000.00 Kz per month and per relative with 4 or more people living in the same household by the end of the study. It will be delivered a total of 11,000.00 Kz per month and per relative with 3 or fewer people living in the same household by the end of the study. The monetary value will be delivered in cash with unconditional format, and it will not be determined by the investigator team the use and the destination of said amount and nothing will be requested in return.
  Interventions: Behavioral: Money transfers

INTERVENTIONS:
Dietary Supplement: Nutritional Supplementation — The Small-quantity lipid-based nutrient supplementation (SQ-LNS) consists of micronutrients delivered in a lipid-based vehicle. All pregnant women (as of 12 weeks self-referred) within households who were randomly included in the study in the nutritional supplementation arm and their children as of 6 months of age will receive the SQ-LNS.
  ● Pregnant women: 20-g sachets, 20 g (1 sachet) dose per day. Nutritional composition and caloric intake.
  Total = 12/13 months approximately.
  ● Children from 6 months of age: 20-g sachets, 20 g (1 sachet) dose per day. Nutritional composition and caloric intake. Total = 18 months.
  The distribution will be made by ADECOS on a fortnightly basis.
  A family ration will be distributed: family supplementation is presented in a basket of locally produced basic foods that complement the usual diet. The caloric distribution of the basket will be 45% of cereals, 30% of pulses, and 25% in oil, and 1 kg of iodized salt.
  Arms: Standard Intervention plus nutritional supplementation (Standard+NUT Arm)
Behavioral: Money transfers — The distribution of the amounts will be made through the corresponding financial providers, together with the Municipal or Communal Administration authorities, the Assistants of Community Activities, the Investigator's personnel, and the ADECOS. The distribution frequency will be every 3 months until the end of the study.
  Arms: Standard Intervention plus money transfers (Standard+TM Arm)
Behavioral: Standard intervention — The activities included are the following:
  1. Community interventions against malnutrition and promotion of adequate nutrition: raise awareness of malnutrition and training mothers to recognize signs of malnutrition.
  2. Community interventions in promoting hygiene and proper sanitation: a) Promotion of Community-Led Total Sanitation approach (CLTS)strategy: community awareness of the entire population included in the cluster about the dangers of open defecation, and the direct link to malnutrition; b) Promotion of Baby-Wash strategy: to make the community aware of the problems and consequences of unsafe water consumption.
  3. Biannual supplementation with vitamin A for children from 6 to 24 months of age.
  4. Biannual deworming (albendazole/mebendazole) for children from 12 months to 24 months of age and pregnant women as of 2nd quarter.
  5. Malaria prophylaxis with sulfadoxine-pyrimethamine (SP) in pregnant women as of 13 weeks of pregnancy.
  Arms: Standard Intervention

SUMMARY:
The severity of the stunting in the provinces of Huíla and Cunene, Angola, in children aged 6 to 59 months is considered to be very high, as defined by the World Health Organization (WHO) classification of 2018. Some of the strategies that present promising results in the fight against chronic malnutrition have been specific nutritional interventions and money transfers. Among these, those that have so far had a greater impact in reducing chronic malnutrition indicators are fortified foods and lipid-based nutrient supplementation in small amounts.

The hypothesis of the study is that these interventions applied from pregnancy can significantly reduce chronic malnutrition, each of which may have different impacts.

The study intends, therefore, to evaluate an intervention that aims to obtain the highest quality scientific evidence on the best package of sensitive and specific measures that reduce chronic malnutrition and mortality in children under 2 years of age, maintaining the fundamental premises of sustainability, cost-benefit ratio, and scalability for other regions of the country.

To this end, it was designed a community trial randomized by clusters in which different strategies will be evaluated separately:

* Standard Intervention The Standard package includes a series of actions carried out by Community and Health Development Agents (ADECOS), which are characterized by having demonstrated strong evidence of their effectiveness in the scientific literature, and are part of the WHO guidelines and national health guidelines in different countries, including Angola.
* Standard+ NUT (Nutrients Arm - Control Arm): Standard Intervention plus nutritional supplementation
* Standard+ TM (Money transfers Arm): Standard Intervention plus money transfers

Study population: pregnant women with more than 16 years of age; however the target population of the interventions will be the household where the pregnant woman lives. The impacts of interventions on indicators of chronic malnutrition in children under 5 years of age belonging to the household will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women of 16 years of age or older;
* Pregnancy confirmed through a test;
* Accept to participate in the study upon the informed consent form is signed by the community leader and confirmed by potential participants.

Exclusion Criteria:

* Women of 16 years of age or older, pregnant, who do not belong to the pre-selected districts/villages of the study;
* Women that, although in the household, are maids, reside in rented homes or are temporary visits;
* Women who have planned to travel or move outside of the district within the study follow-up period;
* Women who manifest the impossibility of completing follow-up visits;
* Alcohol-dependent women or with a history of alcohol abuse (considered as intake of >3 drinks on any day or >7 drinks per week);
* Any condition that, at the investigator's discretion, is non-compliant with interventions or follow-up controls;
* Pregnant women with acute malnutrition (brachial circumference < 21 cm).

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1423 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
● Proportion of children with moderate an serious chronic malnutrition (indices below -2 and -3 Z- scores below the reference median) at 24 months of age in the provinces of Huíla and Cunene. | 24 months
  Effectiveness of three interventions (standard care, money transfers, and nutritional supplements) to reduce chronic malnutrition in children under two years of age in the provinces of Huíla and Cunene by the proportion of children with different degrees of malnutrition.

SECONDARY OUTCOMES:
● Proportion of children under 5 years of age with moderate and severe chronic malnutrition (indices below -2 and -3 Z-scores below the reference median) at the beginning and end of the study in the provinces of Huíla and Cunene. | 0-1 and 24 months
  Effectiveness of three interventions (standard care, money transfers, and nutritional supplements) individually to reduce chronic malnutrition in children under 5 years of age in the provinces of Huíla and Cunene will be assessed by measuring height/length per age score.
Mortality rate at 3, 6, 12, 18, and 24 months after enrollment in the study. | 3, 6, 12, 18, and 24 months
  Mortality will be assessed during all study at selected time frames
Incidence rate in relevant comorbidities | 6, 12, 18, and 24 months
  Incidence of malaria, pneumonia, diarrhea, and anemia (Hemoglobin < 12g/dL) in children up to 2 years of age in the provinces of Huíla and Cunene will be measured.
Increment of food diversity grade at the end of the study compared to baseline. | 0-1 and 24 months
  Attitudes and eating habits of families in the provinces of Huíla and Cunene will be quantified.
Number of pre- and post-natal visits. | 6 months
  Pre- and post-natal care indicators such as exclusive breastfeeding rate in children up to 6 months of age and low birth weight will be assessed
Cost-effectiveness incremental ratios (obtained dividing the incremental cost by the incremental benefit for health ). | 2 years
  The cost-effectiveness of different interventions will be measured.
Proportion of children with moderate and severe chronic malnutrition (indices below -2 and -3 Z- scores below the reference median) at 3, 6, 12, 18, months of age in the provinces of Huíla and Cunene. | 3, 6, 12, 18 months
  Effectiveness of three interventions (standard care, money transfers, and nutritional supplements) to reduce chronic malnutrition in children under two years of age in the provinces of Huíla and Cunene by the proportion of children with different degrees of malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Molina, Study Chair — Vall d'Hebron Institut de Recerca (VHIR)
Locations (2):
- Angola (2):
  - Cunene, Otchinjau; Mupa, Cunene Province
  - Huíla province, Libongue; Jamba Sede

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin-Canavate R, Trigo E, Romay-Barja M, Faria LM, Gerardo AS, Aguado I, Iraizoz E, Marques T, Molina I, Custodio E. Dietary Diversity in Pregnant Women and Its Association With Household Food Security in Rural Southern Angola. Matern Child Nutr. 2025 Oct;21(4):e70051. doi: 10.1111/mcn.70051. Epub 2025 Jun 2. PMID 40457576
- [Derived] Custodio E, Herrador Z, Trigo E, Romay-Barja M, Ramirez F, Aguado I, Iraizoz E, Silva-Gerardo A, Faria ML, Martin-Canavate R, Marques T, Vargas A, Gomez A, Molina I. Nutrition supplementation plus standard of care versus standard of care alone or standard of care plus unconditional cash transfer in the prevention of chronic malnutrition in Southern Angola: study protocol for the MuCCUA study, a cluster randomized controlled trial. BMC Public Health. 2024 Feb 10;24(1):429. doi: 10.1186/s12889-024-17858-7. PMID 38341528
- [Derived] Martin-Canavate R, Custodio E, Trigo E, Romay-Barja M, Herrador Z, Aguado I, Ramirez F, Faria LM, Silva-Gerardo A, Lima JC, Iraizoz E, Marques T, Vargas A, Gomez A, Puett C, Molina I. Preventing chronic malnutrition in children under 2 years in rural Angola (MuCCUA trial): protocol for the economic evaluation of a three-arm community cluster randomised controlled trial. BMJ Open. 2023 Dec 18;13(12):e073349. doi: 10.1136/bmjopen-2023-073349. PMID 38110392
- See also: Operational research against chronic child malnutrition in Angola (CRESCER Project) — https://crescerangola.com/